CLINICAL TRIAL: NCT00636545
Title: A Safety, Pharmacokinetic, and Pharmacodynamic Assessment of Genasense Administered as a 2-hour Intravenous Infusion to Subjects With Solid Tumors
Brief Title: Genasense as a 2-hour Intravenous Infusion in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPK109
Record Dates: First submitted 2007-10-11; First posted 2008-03-14 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2009-01

CONDITIONS: Solid Tumors
Keywords: Genasense; oblimersen; antisense; Bcl-2 antisense; Solid Tumors
MeSH Terms: interventions — oblimersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Cohort 1- Genasense will be administered as a 2-hour intravenous infusion once weekly for 3 weeks at a dose of 300 mg to the first subject enrolled and, in the absence of dose-limiting toxicity, in increasing increments of 100 mg to each successive subject enrolled to a maximum dose of 1000 mg.
  Interventions: Drug: Oblimersen (Genasense)
- Part 2 (Experimental): Genasense will be administered as a 2-hour intravenous infusion twice weekly for 3 weeks at a dose established based on Part 1 of the study.
  Interventions: Drug: Oblimersen (Genasense)
- Cohort 2 (Experimental): Also in Part 1 of the study, Genasense will be administered as a 2-hour intravenous infusion once weekly for 3 weeks at a starting dose of 1100 mg and increasing in increments of 100 mg to the MTD. Patients will be pretreated with a corticosteroid.
  Interventions: Drug: Oblimersen (Genasense)

INTERVENTIONS:
Drug: Oblimersen (Genasense) — Intravenous
  Other Names: Oblimersen; Oblimersen sodium; Genasense; G3139; Bcl-2 antisense oligonucleotide
  Arms: Part 1; Part 2
Drug: Oblimersen (Genasense) — Intravenous
  Arms: Cohort 2

SUMMARY:
The primary objective is to determine the safety and maximum tolerated dose (MTD) of Genasense administered as a 2-hour intravenous infusion once weekly (Part 1) and twice weekly (Part 2) to patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a solid tumor malignancy, not to include lymphoma, that has failed standard therapy or for which no standard therapy is available
* Adequate organ function as determined ≤ 7 days prior to starting study medication
* Eastern Cooperative Oncology Group performance status 0 to 2
* At least 3 weeks and recovery from effects of major prior surgery or other therapy, including chemotherapy, radiation therapy, immunotherapy, or cytokine, biologic, or vaccine therapy

Exclusion criteria

* Other significant medical disease
* History or presence of leptomeningeal disease
* Coexisting condition that would require the subject to continue therapy during the treatment phase of the study with a drug known to alter renal function
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Genasense administered as a 2-hour IV infusion once a week (Part 1) and twice a week (Part 2) to patients with solid tumors | One year

SECONDARY OUTCOMES:
Pharmacokinetics (Part 1 and Part 2); pharmacodynamics (Part 2) | During treatment phase

CONTACTS AND LOCATIONS:
Locations (1):
- South Texas Accelerated Research Therapeutics, San Antonio, Texas, United States